CLINICAL TRIAL: NCT07382128
Title: Myocardial Perfusion CMR for Differentiating and Characterizing Hypertrophic Cardiomyopathy Phenotypes
Acronym: MyoPerf-HCM
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: MyoPerf-HCM
Record Dates: First submitted 2026-01-26; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: HCM - Hypertrophic Cardiomyopathy; Anderson Fabry Disease; Cardiac Magnetic Resonance Imaging; Amyloid Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Fabry Disease; Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to evaluate myocardial perfusion abnormalities using quantitative and qualitative cardiac magnetic resonance (CMR) perfusion imaging in patients with hypertrophic cardiomyopathy (HCM) phenotypes, including sarcomeric and non-sarcomeric HCM, Anderson-Fabry disease (AFD), and cardiac amyloidosis. The study will also include first-degree relatives of affected patients and genetic mutation carriers. By comparing myocardial blood flow and perfusion patterns across these different conditions, the study seeks to identify distinctive perfusion signatures that may improve diagnostic differentiation, support risk stratification, and provide insights into the role of ischemia in fibrosis progression, arrhythmias, and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of cardiomyopathy with a hypertrophic phenotype, according to current ESC guidelines; or a first-degree relative of a patient with a confirmed diagnosis of cardiomyopathy with a hypertrophic phenotype; or a carrier of a genetic mutation for hypertrophic cardiomyopathy (carriers).
* Patient with an indication to undergo cardiac magnetic resonance imaging (CMR) according to current ESC guidelines.
* Age ≥ 18 years
* Written informed consent obtained

Exclusion Criteria:

- History of previous myocardial infarction or myocardial revascularization (coronary artery bypass grafting or percutaneous coronary angioplasty) and/or evidence of coronary stenosis ≥ 50% on coronary CT scan or invasive coronary angiography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients will participate in the study, including those with a confirmed diagnosis of hypertrophic-phenotype cardiomyopathies (sarcomeric and non-sarcomeric HCM, Anderson-Fabry disease, amyloidosis), first-degree relatives of patients with a confirmed diagnosis of hypertrophic-phenotype cardiomyopathy, and carriers of genetic mutations associated with hypertrophic cardiomyopathy.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative Perfusion Defects | Baseline and after 36 months
  To evaluate differences in quantitative myocardial perfusion among different hypertrophic cardiomyopathy phenotypes, aiming to identify specific and distinctive perfusion abnormality patterns for each condition.
Qualitative Perfusion Defects | Baseline and after 36 months
  To evaluate differences in qualitative myocardial perfusion among different hypertrophic cardiomyopathy phenotypes, aiming to identify specific and distinctive perfusion abnormality patterns for each condition.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No